CLINICAL TRIAL: NCT04123951
Title: A Pilot Randomised Controlled Trial of the Effects of a Structured, Home-based Exercise Program on Cardiovascular StructurE and Function in Renal Transplant Recipients: The ECSERT Study
Brief Title: Home-based Exercise in Renal Transplant Recipients
Acronym: ECSERT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0714
Record Dates: First submitted 2019-09-16; First posted 2019-10-11 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant; Complications
Keywords: Kidney Transplant; Cardiovascular Disease; Home-based Exercise; Exercise
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Exercise (Experimental): Patients in this arm will complete a 12 week home-based aerobic and resistance exercise training programme. There will be a 2 week period prior to this in which patients will complete up to 6 supervised sessions in order to learn about the home-based exercise training. There will be a 4 week return visit and an optional 8 week return visit in order to reassess fitness and aid the patients with any questions or queries they may have and to aid them in progressing their exercise.
  Interventions: Other: Home-based Exercise
- Control (No Intervention): In this arm patients will continue 'as normal' with daily activities.
  Patients in this arm will be offered the exercise intervention once they have completed post 12 week assessments.

INTERVENTIONS:
Other: Home-based Exercise — Patients in the home-based exercise arm will complete a 12 week home-based aerobic and resistance exercise training programme. There will be a 2 week period prior to this in which patients will complete up to 6 supervised sessions in order to learn about the home-based exercise training. There will be a 4 week return visit and an optional 8 week return visit in order to reassess fitness and aid the patients with any questions or queries they may have and to aid them in progressing their exercise.
  Arms: Home-based Exercise

SUMMARY:
Although patients who have received a kidney transplant have better health than patients on dialysis, heart problems are still the commonest cause of death for kidney transplant recipients. This is because diseases like high blood pressure and diabetes are more common in patients with kidney transplants as well as factors related to having kidney disease itself and the medications transplant recipients have to take to stop them rejecting their transplanted kidney. Exercise is known to help with heart disease in lots of conditions and improves many of the risk factors known to cause heart disease in kidney transplant recipients. This study will investigate whether an individualised, home-based, exercise program improves heart disease in kidney transplant recipients. The study is a randomised controlled trial, with half the patients completing the 12 week exercise programme and the other half continuing with their normal care. The investigators will use detailed MRI scans to assess patient's hearts and blood vessels at the start and end of the study. The investigators will also assess changes in physical function, exercise capacity, blood markers of heart disease, changes in body type and quality of life measures assessed with questionnaires.

DETAILED DESCRIPTION:
Kidney transplantation confers a significant survival advantage over remaining on dialysis, but CVD remains the leading cause of death for RTRs and of graft loss. Acute myocardial infarction accounts for 15-20% of CVD-related deaths in RTRs, but sudden cardiac death, or death from fatal arrhythmia account for at least double this number, suggesting classical atheromatous coronary artery disease driven by traditional cardiometabolic risk factors, is not the dominant driving force of CVD in RTRs. Non-traditional cardiometabolic risk factors including endothelial dysfunction, systemic inflammation, acute rejection, anaemia and deranged bone-mineral metabolism are of at least equal importance in the pathogenesis of CVD in RTRs and drive pathological changes in cardiovascular structure and function that associate strongly with mortality. This is further illustrated by the fact that traditional CVD risk-stratification tools dramatically underestimate cardiovascular risk in patients with CKD, coronary revascularization does not improve outcomes for RTRs as it does in the general population and cardiac events are more likely to be fatal in RTRs than the general population. Immunosuppressive agents are well known to drive traditional CVD risk factors, but also drive non-traditional cardiometabolic risk factors. Cost-effective, deliverable interventions are needed to address the burden of CVD in RTRs by targeting traditional and non-traditional risk factors. Supervised exercise interventions in RTRs improve cardiorespiratory fitness and a variety of traditional and non-traditional risk factors for CVD, including metabolic profile, vascular stiffening, central adiposity and inflammatory cell and cytokine profiles, but are not realistically deliverable in the current financial climate. Home-based exercise training programs have been shown to be deliverable in patients on dialysis and patients undergoing cardiac rehabilitation, but the effectiveness and deliverability of home-based exercise interventions are largely untested in RTRs. It cannot be assumed such programs will be acceptable to RTRs, whose home-lives, social and occupational circumstances are significantly different to dialysis and cardiac patients. Many RTRs have had enforced sedentary lifestyles prior to transplantation as dialysis patients and their goals for rehabilitation as well as the disease processes at work are different to both dialysis and cardiac patients.

There are limited data on whether exercise-induced improvements in cardiometabolic risk translate into improvements in cardiovascular structure and function in RTRs. CMR is able to measure multiple clinically pertinent aspects of CVD processes in RTRs that relate closely to outcome with great accuracy, including:

* left ventricular hypertrophy
* myocardial fibrosis
* aortic stiffness
* coronary artery function
* myocardial steatosis
* subclinical systolic and diastolic dysfunction

This pilot randomised clinical trial will assess the deliverability of a combined aerobic and resistance, home-based, exercise intervention in RTRs. It will define recruitment and dropout rates from this newly designed, home-based, intervention and baseline values for CMR measures that assess prognostically important aspects of CVD in RTRs for the first time. Furthermore, it will test the effects of the intervention on traditional and novel CMR outcome measures that assess prognostically important aspects of CVD that relate directly to cardiovascular outcomes for the first time, providing estimates of effect-sizes on outcome measures. These data will be used to inform the design of a future, definitive study. This study will further the investigator's ability to make objective measures of cardiovascular health in RTRs, with the opportunity to compare CMR measures with traditional measures of cardiovascular fitness. The qualitative component of this study will refine the exercise intervention to maximize uptake in future studies and adoption into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age great than 18 years old
* Prevalent RTR longer than 1year
* Able and willing to give informed consent
* Increased cardiometabolic risk, with at least one of:

Diabetes mellitus Dyslipidaemia Hypertension History of ischaemic heart disease or cerebrovascular disease Obesity (BMI above 30)

Exclusion Criteria:

* Unable to undertake exercise due to physical or psychological barriers
* Unable to undergo CMR scanning (incompatible implants, claustrophobia, allergy to agents)
* Contraindication to exercise training (American College of Sports Medicine guidelines)
* Female participants who are pregnant, lactating, or planning pregnancy during the course of the study.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Any other significant disease or disorder (i.e. significant co-morbidity including unstable hypertension, potentially lethal arrhythmia, myocardial infarction within 6 months, unstable angina, active liver disease, uncontrolled diabetes mellitus (HbA1c greater than or equal to 9%), advanced cerebral or peripheral vascular disease) which, in the opinion of the patient's own clinician the Principle Investigator may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Inability to give informed consent or comply with testing and training protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Left ventricular mass (g/m) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)
Change in left/right ventricular volumes (ml) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)
Change in ejection fractions (%) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)
Change in native and post-contrast T1 mapping time (ms) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)
Change in Myocardial systolic-strain (%) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)
Change in peak early-diastolic strain rate (%s-1) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)
Change in Aortic pulse wave velocity (m/s) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)
Change in aortic distensibility (mmHg-1×10-3) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)
Change in Myocardial and hepatic triglyceride content (%) | Baseline and 12 weeks
  Measured using multi-parametric cardiac MRI (CMR)

SECONDARY OUTCOMES:
Recruitment Rate | Post 12 week intervention
  The feasibility of recruitment and interest of patients is an essential component of whether a full trial is feasible. The number of eligible patients and number of consented will be recorded. Monthly recruitment rate and the time taken to recruit 10 (25%), 20 (50%), 30 (75%), and 40 (100%) patients will be recorded.
Number of participants lost to follow up | Post 12 week intervention
  This is the number of participants leaving the trial due to being uncontactable
Number of exercise sessions completed per week | Post 12 week intervention
  This will assess adherence to the intervention
Number of participants dropping out of the trial | Post 12 week intervention
  Otherwise known as the attrition rate
Number of adverse events | Post 12 week intervention
  This is a measure of the trial safety
Aerobic Capacity (change) | Baseline, 2 weeks, 4 weeks and 12 weeks
  Measured by cardiopulmonary exercise test which produces V02 (maximal oxygen uptake) in both l/min and ml/kg/min. This is a measure of a participants aerobic capacity.
Timed up and go test (TUAG)(change) | Baseline and 12 weeks
  To determine fall risk and measure the progress of balance, sit to stand and walking. Patient sits and then the time taken to stand up and walk 3 meters and return is measured. If a patient took 14 seconds or longer he or she was classified as high-risk for falling
Habitual Physical Activity (change) | Baseline and 12 weeks
  Via accelerometry
Lower limb strength (change) | Baseline and 12 weeks
  Dynamometry
Upper Limb Strength (change) | Baseline and 12 weeks
  Hand grip
Change in circulation markers of systemic inflammation | Baseline and 12 weeks
  Blood Sampling including but not limited to IL-6, CRP, IL-10, TNF-Alpha
Muscle quality using Ultrasound Imaging (change) | Baseline and 12 weeks
  Cross-sectional area (cm2)
Muscle quality using Ultrasound Imaging (change) | Baseline and 12 weeks
  fat thickness (mm)
Muscle Elasticity (change) | Baseline and 12 weeks
  Muscle elasticity will be measures using a MyotonPro device
Lower limb endurance (change) | Baseline and 12 weeks
  Sit to stand 60 test measuring how many 'sit to stands' can be performed in 60 seconds
Balance (change) | Baseline and 12 weeks
  Measured using a 'wii-fit' style board. Better balance is an idicator of falls risk
Gait speed (change) | Baseline and 12 weeks
  Gait speed is measure as the time taken to walk 4 meters. Slower speeds have been linked to higher mortality risk
Height | Baseline
  Height measured in meters
Weight (change) | Baseline and 12 weeks
  Weight measured in kg
Body fat % (change) | Baseline and 12 weeks
  Body fat measured using bio electrical impedance analysis

OTHER OUTCOMES:
Integrated Palliative care Outcome Scale for Renal (I-POS-Renal)(change) | Baseline and 12 weeks
  IPOS-Renal is a short measure (11 questions), combining the most common symptoms renal patients experience plus additional items from IPOS on concerns beyond symptoms, such as information needs, practical issues, family anxiety. IPOS has been validated in a mixed population of those with cancer and non-cancer diagnosis, including renal patients, and shows good content and construct validity, reliability, and responsiveness to change. Each symptom is rated on a scale of 0-4 for how much that symptom effects the participant. 0 is not at all and 4 is severely. Higher total scores indicate more symptom burden.
Short Form Health Survey (SF-12)(change) | Baseline and 12 weeks
  Categorical questions that assess limitations in role functioning as a result of physical and emotional health. The survey also contains Likert response formats including those that are on a three-point scale (e.g., limited a lot, limited a little, or not limited at all) that assess limitations in physical activity and physical role functioning. A five-point scale (e.g., not at all, a little bit, moderately, quite a bit, and extremely) that assesses pain, and a five-point scale that assesses overall health (excellent, very good, good, fair, and poor) are included. The SF-12 also contains a six-point scale (e.g., all of the time, most of the time, a good bit of the time, some of the time, a little of the time, and none of the time) that assesses mental health, vitality, and social functioning. Two summary scores: mental health (MCS12), and physical health (PCS12). The scores are represented as t-scores that are linear transformations with a mean of 50 and a standard deviation of 10
Patient Activation Measure (PAM)(Change) | Baseline and 12 weeks
  Individuals are asked to complete a short survey and based on their responses, they receive a PAM score (between 0 and 100). The resulting score places the individual at one of four levels of activation, each of which reveals insight into a range of health-related characteristics, including behaviours and outcomes. The four levels of activation are:
  Level 1: Individuals tend to be passive and feel overwhelmed by managing their own health. They may not understand their role in the care process.
  Level 2: Individuals may lack the knowledge and confidence to manage their health.
  Level 3: Individuals appear to be taking action but may still lack the confidence and skill to support their behaviours.
  Level 4: Individuals have adopted many of the behaviours needed to support their health but may not be able to maintain them in the face of life stressors.
  Particulars of the scoring system (and scales) are not disclosed by the license holder
(FACIT-F)(change) | Baseline and 12 weeks
  The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue with a 7-day recall period. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue
Pittsburgh Sleep Quality Index (PSQI)(change) | Baseline and 12 weeks
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Graham-Brown, Principal Investigator — University of Leicester
Locations (1):
- University Hospital Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Billany RE, Vadaszy N, Burns S, Chowdhury R, Ford EC, Mubaarak Z, Sohansoha GK, Yeo JL, Dattani A, Cowley AC, Gulsin GS, Bishop NC, Smith AC, McCann GP, Graham-Brown MP. Cardiorespiratory fitness in kidney transplant recipients: A pilot randomised controlled trial of structured home-based rehabilitation and a nested case-control analysis. Clin Rehabil. 2025 Dec 30:2692155251408792. doi: 10.1177/02692155251408792. Online ahead of print. PMID 41468011
- [Derived] Billany RE, Macdonald JH, Burns S, Chowdhury R, Ford EC, Mubaarak Z, Sohansoha GK, Vadaszy N, Young HML, Bishop NC, Smith AC, Graham-Brown MPM. A structured, home-based exercise programme in kidney transplant recipients (ECSERT): A randomised controlled feasibility study. PLoS One. 2025 Feb 24;20(2):e0316031. doi: 10.1371/journal.pone.0316031. eCollection 2025. PMID 39992959
- [Derived] Billany RE, Vadaszy N, Bishop NC, Wilkinson TJ, Adenwalla SF, Robinson KA, Croker K, Brady EM, Wormleighton JV, Parke KS, Cooper NJ, Webster AC, Barratt J, McCann GP, Burton JO, Smith AC, Graham-Brown MP. A pilot randomised controlled trial of a structured, home-based exercise programme on cardiovascular structure and function in kidney transplant recipients: the ECSERT study design and methods. BMJ Open. 2021 Oct 5;11(10):e046945. doi: 10.1136/bmjopen-2020-046945. PMID 34610929